CLINICAL TRIAL: NCT00616512
Title: A Randomized Controlled Trial of a Water Protocol for Clients With Thin Liquid Dysphagia: a Pilot Project
Brief Title: A Randomized Controlled Trial of a Water Protocol for Clients With Thin Liquid Dysphagia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: B.C. Rehabilitation Foundation (Other)
Responsible Party: Caren Carlaw, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H07-02582
Record Dates: First submitted 2008-02-04; First posted 2008-02-15 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: Thin Liquid Dysphagia
Keywords: Water; oral care; oral hygiene; dysphagia; thin liquid dysphagia; thickened liquids
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): GF Strong Water Protocol/ water allowed between meals after oral care for selected clients/ Fraser Water Protocol
  Interventions: Procedure: GF Strong Water Protocol

INTERVENTIONS:
Procedure: GF Strong Water Protocol — The Purpose of the GF Strong water protocol is to allow clients who have thin liquid dysphagia to drink water under certain specified conditions according to the rules of the water protocol.

SUMMARY:
The Purpose of the GF Strong water protocol is to allow clients who have thin liquid dysphagia to drink water under certain specified conditions according to the rules of the water protocol. Water Protocols have been shown to improve client satisfaction, and hydration. We wish to assess this in a randomized, controlled fashion, and this is a pilot project to determine feasibility.

DETAILED DESCRIPTION:
GF Strong water protocol will be used with the study subjects. Control subjects will not receive water protocol. Pre and post measures will include SWAL-QOL, client satisfaction, water and thickened fluid intake, and monitoring for adverse events.

ELIGIBILITY:
Inclusion Criteria:

Potential participants in this study will include all clients aged 19 years and older who are admitted to GF Strong Acquired Brain Injury (ABI) and Neruomusculoskeletal (NMS) and Adolescent and Young Adult (AYA) programs and who have thin liquid dysphagia resulting from a neurological diagnosis. The thin liquid dysphagia will be confirmed by a Modified Barium Swallow conducted by a certified speech-language pathologist. Potential participants must be proficient in English in order to complete the questionnaires and capable of understanding the consent form.

Exclusion Criteria:

Clients who present with the following will be excluded: active pneumonia, acute or unstable medical condition, surgery where coughing might rip stitches or cause pain or discomfort, oral dental bacteria or infection that cannot be controlled, poor oral hygiene that cannot be improved with routine care, excessive or uncomfortable coughing during or after intake, severe or uncontrolled GERD, immunosuppressed, or decline participation.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-04; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Feasibility | Information not available

SECONDARY OUTCOMES:
Fluid intake, client satisfaction, quality of life, adverse events | Information not available

CONTACTS AND LOCATIONS:
Overall Officials: Caren Carlaw, MA, Principal Investigator — University of British Columbia; Heather Finlayson, MD, FRCPC, Study Director — University of British Columbia; Kathleen Beggs, Bse RDN, Study Director — University of British Columbia; Andrew Travlos, MBBCh FRCPC, Study Director — University of British Columbia; Dawn Coney, RN (CRN), Study Director — University of British Columbia; Tiffany Visser, MS, Study Director — University of British Columbia; Caroline Marcoux, MS, Study Director — University of British Columbia
Locations (1):
- GF Strong Rehabilitation Centre, Vancouver, British Columbia, Canada